CLINICAL TRIAL: NCT00636129
Title: Biochemical and Physiological Changes Associated With Differing Durations of Relaxation Response Training
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Herbert Benson, Director Emeritus, Benson-Henry Institute for Mind Body Medicine, Massachusetts General Hospital
Other Study IDs: MIT COUHES 577
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Stress
Keywords: relaxation; relaxation response; meditation; nitric oxide; stress management; stress; Relaxation Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Relaxation Response + Stress Management Curriculum
  Interventions: Behavioral: Relaxation Response + Stress Management Curriculum

INTERVENTIONS:
Behavioral: Relaxation Response + Stress Management Curriculum — Subjects will receive 8 weeks of Stress Management curriculum and guidance through 20 minute Relaxation Response with a research coordinator. They will also practice 20 minutes of Relaxation Response at home daily.

SUMMARY:
We are looking at the effects of Stress Management and Relaxation Response training on stress hormones (like adrenalin and cortisol), immune function and physiology (heart rate, breathing rate, muscle tension).

DETAILED DESCRIPTION:
The primary aim of this study is to determine whether differing durations of relaxation response (RR) training will be associated with different degrees of change in physiological, psychological, hormonal, molecular and immunological markers. Prior studies have reported reduction on many of these parameters after 8 weeks of RR training. However, we now seek to understand the degree to which incremental decreases in these parameters are exhibited at 0, 4, and 8 weeks of RR practice in 30 healthy adults. Furthermore, we will explore correlations between levels of exhaled nitric oxide or plasma nitrites/nitrates and oxygen consumption during RR elicitation. We will also examine any associations between changes in oxygen consumption and psychological factors, physiological parameters, and biochemical outcomes. Lastly, we will bank plasma and peripheral blood cells from these samples for future assessments of immune markers, cell typing and gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49
* Healthy subjects

Exclusion Criteria:

* Taking medication
* Asthma or allergies
* Prior regular relaxation practice
* Body Mass Index >39
* Beck Depression Inventory (BDI) score indicates possible clinical depression
* Current mental health treatment
* Diagnosis of severe mental illness
* Using hormonal birth control
* Females: pregnant or trying to conceive
* Exhaled Nitric Oxide (NO) levels > 60PPB
* Hematocrit < 32%
* Blood glucose < 50 or > 200
* Creatinine > 1.3

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects ages 18-49.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Benson, MD, Principal Investigator — Benson-Henry Institute for Mind Body Medicine at Massachusetts General Hosptial
Locations (1):
- Benson-Henry Institute for Mind Body Medicine, Boston, Massachusetts, United States